CLINICAL TRIAL: NCT04027868
Title: Cohort Study to Evaluate the Clinical Features of Patients With Epithelial Ovarian Cancer Depending on Tumoral Mutation of BRCA or Beyond BRCA Genomic Molecular Abnormalities
Brief Title: Genomic BRCA and Extensive ovArian Cancer Testing
Acronym: GREAT
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: GINECO-OV128; 2019-A01190-57 (Other: ANSM); 19.06.45 (Other: Ethics Committee)
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tumor sample fixed in formalin and included in paraffin (FFPE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational French multicenter cohort in patients with ovarian and/or primitive peritoneal and/or fallopian tubes carcinoma, histologically confirmed, with an advanced stage at diagnosis (stage III to IV FIGO 2014). The objective is to constitute a clinico-biological database that allows to correlate clinical and progressive features of ovarian cancer patients based on tumor genomics and molecular detected abnormalities.

DETAILED DESCRIPTION:
This is a prospective observational French multicenter cohort in patients with ovarian and/or primitive peritoneal and/or fallopian tubes carcinoma, histologically confirmed, with an advanced stage at diagnosis (stage III to IV FIGO 2014). The objective is to constitute a clinico-biological database that allows to correlate clinical and progressive features of ovarian cancer patients based on tumor genomics and molecular detected abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Patient with ovarian and/or primitive peritoneal and/or fallopian tubes carcinoma, histologically confirmed, with an advanced stage at diagnosis (stage III to IV FIGO 2014)
* Patient in first line therapy
* Available tumor sample fixed in formalin and included in paraffin (FFPE):

  * in pre-chemotherapy, insofar as possible
  * having a sufficient tumor surface, with a final cellularity of at least 20%
* Identification of a molecular genetics' cancer platform participant in GREAT and an onco-geneticists team working with the investigator team
* Patient consenting her data to be collected and submitted through an automated processing
* Patient beneficiary from the French social security

Exclusion Criteria:

* Patient with a mucinous ovarian carcinoma
* Patient pregnant or breastfeeding
* Patient under legal protection (guardianship or court order) or unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian and/or primitive peritoneal and/or fallopian tubes carcinoma, histologically confirmed, with an advanced stage at diagnosis (stage III to IV FIGO 2014)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Correlation between Progression Free Survival (PFS) and the detected tumor genetic abnormalities | From baseline until the date of progression or death, which ever occurs earlier, assessed up to 10 years

SECONDARY OUTCOMES:
Correlation between age and the detected tumor genetic abnormalities | Baseline
Correlation between histology status and the detected tumor genetic abnormalities | Baseline
Correlation between FIGO stage and the detected tumor genetic abnormalities | Baseline
Correlation between surgery resection status and the detected tumor genetic abnormalities | Up to 10 years
Correlation between treatment response and the detected tumor genetic abnormalities | Up to 10 years
Correlation between Overall survival (OS) and the detected tumor genetic abnormalities | From baseline to death, assessed up to 10 years

OTHER OUTCOMES:
Percentage of patients with both germinal and tumoral BRCA tests | Up to 10 years
Percentage of patients with a first germinal BRCA test, a first tumoral BRCA test, or simultaneous germinal and tumoral tests | Up to 10 years
Percentage of patients with and exploitable tumoral block for exploratory transversal researches | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Thibault De La Motte Rouge, MD., Principal Investigator — Centre Eugène Marquis, Rennes
Locations (137):
- France (137):
  - Centre de Radiothérapie et d'Oncologie de Moyenne Garonne (CROMG), Agen
  - Hôpital Privé d'Aix en Provence, Aix-en-Provence
  - Centre Hospitalier Général d'Aix-en-Provence, Aix-en-Provence
  - CHU Amiens, Amiens
  - Clinique Victor PAUCHET, Amiens
  - Institut de Cancérologie de l'Ouest - ICO, Angers
  - Hôpital Privé d'Antony - Ramsay Santé, Antony
  - CH Arras, Arras
  - CH Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Clinique Belharra, Bayonne
  - CH Côte Basque, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - CHRU Jean Minjoz, Besançon
  - Reims Icone, Bezannes
  - CH de Blois, Blois
  - Hôpital Avicenne, Bobigny
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Hospitalier Fleyriat - BOURG-EN-BRESSE, Bourg-en-Bresse
  - CHU Brest, Brest
  - Hôpital Femme Mère Enfant, Bron
  - Centre François Baclesse, Caen
  - Centre Maurice Tubiana, Caen
  - CH de Cahors, Cahors
  - CH Carcassonne, Carcassonne
  - Hôpital Général de Castres, Castres
  - Medipole de Savoie, Challes-les-Eaux
  - CH Chalon sur Saone, Chalon-sur-Saône
  - CH Metropole Savoie, Chambéry
  - Centre d'Oncologie et de Radiothérapie 37, Chambray-lès-Tours
  - Centre Hospitalier de Chateauroux, Châteauroux
  - CHPC - Hôpital Louis Pasteur, Cherbourg
  - CH Cholet, Cholet
  - Hôpital Antoine Béclère, Clamart
  - Centre Jean Perrin, Clermont-Ferrand
  - CH Alpes Léman, Contamine-sur-Arve
  - Centre Hospitalier Sud Francilien (Site Gilles de Corbeil), Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - Clinique de Flandre, Coudekerque-Branche
  - Groupe Hospitalier public du Sud de l'Oise (GHPSO), Creil
  - CHI Creteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU Dijon, Dijon
  - Institut de Cancérologie de Bourgogne - GRReCC, Dijon
  - Clinique du Mousseau (CMCO) - Ramsay Santé, Évry
  - Centre Hospitalier Intercommunal de Fréjus Saint Raphael, Fréjus
  - GH Mutualiste de Grenoble, Grenoble
  - Hôpital Privé Drôme Ardèche - Clinique Pasteur, Guilherand-Granges
  - Centre Hospitalier Marne-la-Vallée, Jossigny
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - CHU Grenoble Alpes - Site Nord (La Tronche), La Tronche
  - Hôpital André Mignot, Le Chesnay
  - Les Hôpitaux de Chartres, Le Coudray
  - Hôpital Privé de l'Estuaire, Le Havre
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier du Mans, Le Mans
  - CH de Lens, Lens
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Polyclinique de Limoges - Clinique Chenieux, Limoges
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Groupe Hospitalier Bretagne Sud - Hôpital du Scorff, Lorient
  - HCL - Hôpital de la Croix Rousse, Lyon
  - Clinique de l'infirmerie Protestante, Lyon
  - Centre Léon Bérard, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - APHM - Hôpital de la Timone, Marseille
  - Hôpital Nord, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Layné, Mont-de-Marsan
  - Hôpital Nord Franche Comté, Montbéliard
  - CH de Montelimar, Montélimar
  - Centre de Cancérologe du Grand Montpellier, Montpellier
  - CHRU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - ICM - Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Oracle - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancérologie du Gard - ONCOGARD, Nîmes
  - Institut de Cancérologie du Gard, Nîmes
  - CHR Orléans, Orléans
  - Hôpital de la Pitié Salpétrière, Paris
  - GH Saint Joseph, Paris
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - HEGP, Paris
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Lariboisière, Paris
  - Institut Curie, Paris
  - Institut Mutualiste Montsouris, Paris
  - CH Pau, Pau
  - Centre Catalan d'Oncologie, Perpignan
  - CH Perpignan, Perpignan
  - Clinique Francheville, Périgueux
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO-HPCA, Plérin
  - Hôpital de la Milétrie, Poitiers
  - CH René Dubos, Pontoise
  - CH Annecy Genevois, Pringy
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Centre Eugène Marquis, Rennes
  - Hôpitaux Drôme Nord - Centre Hospitalier Romans, Romans-sur-Isère
  - Centre Henri Becquerel, Rouen
  - Clinique Mathilde, Rouen
  - Centre Frédéric Joliot, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Institut Curie - Site Saint Cloud, Saint-Cloud
  - Hôpital Privé de La Loire Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest - ICO, Saint-Herblain
  - HIA Begin, Saint-Mandé
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - Centre Médicale Sainte Feyre Alfred Leune, Sainte-Feyre
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Institut de Cancérologie Paris Nord, Sarcelles
  - CH Sens, Sens
  - CH Broussais, St-Malo
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hôpital Foch, Suresnes
  - CHR Metz-Thionville / Hôpital de Mercy, Thionville
  - Hôpitaux du Léman, Thonon-les-Bains
  - Hôpital d'Instruction des Armées Saint-Anne, Toulon
  - Clinique Pasteur - Groupe Oncorad Garonne, Toulouse
  - Clinique Pasteur - Oncosud, Toulouse
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - Centre Hospitalier de Troyes, Troyes
  - CH Jean Bernard, Valenciennes
  - Clinique des Dentellières, Valenciennes
  - Institut de Cancérologie de Lorraine (ICL) - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No